CLINICAL TRIAL: NCT07224412
Title: Utilizing Digital Health Approaches to Promote Early Childhood Healthy Eating and Activity Behaviors
Brief Title: A Digital Intervention to Promote Preschool Nutrition and Activity: The eHEROs Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB0010703; 2021-68015-34557 (Other Grant/Funding Number: USDA NIFA)
Record Dates: First submitted 2025-10-22; First posted 2025-11-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Health Behavior
Keywords: parents; child, preschool; mHealth; mobile app; nutrition; physical activity
MeSH Terms: conditions — Health Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: parallel pilot feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KnowHow Program (Experimental): Families will participate in the 10-week KnowHow program and will receive/participate in 1) a custom mobile application (app), 2) virtual group discussions, and 3) child-centered support materials
  Interventions: Behavioral: KnowHow Program
- Wait List (No Intervention): Families will not receive any intervention during the 10-week study. Families will receive access to the KnowHow app only for 10 weeks at the conclusion of the study.

INTERVENTIONS:
Behavioral: KnowHow Program — The KnowHow intervention is a 10-week program that provides parent education on the topics of mindful parenting, healthy eating, and physical literacy. The intervention consists of three components: 1) a custom mobile application (app), 2) virtual group discussions, and 3) child-centered support materials mailed to participating families. (1) The KnowHow app will provide parent education using a variety of modalities The 'know' will provide parents with the core information on mindful parenting, healthy eating, and physical literacy, and the 'how' will give strategies to incorporate the information into daily routines and activities. To facilitate the transition from the 'know' to 'how', the app will have a 'Kid Zone' with content to engage in activities with the preschooler. KnowHow app content will be divided into five modules that include A) lessons (text, audio, video), B) activities, and C) assessments. (2) During the 10-week intervention, participants will also meet via Zoom for
  Other Names: eHEROs
  Arms: KnowHow Program

SUMMARY:
The purpose of this pilot study is to assess the feasibility and acceptability of the Know-How program, a 10-week digital intervention for families of young children promoting healthy eating and activity behaviors and environments.

DETAILED DESCRIPTION:
The purpose of this pilot study is to assess the feasibility and acceptability of the KnowHow program, a 10-week digital intervention for families of young children promoting healthy eating and activity behaviors and environments. The KnowHow program, which provides parent education on the topics of mindful parenting, healthy eating, and physical literacy, consists of three components: 1) a custom mobile application (app), 2) virtual group discussions, and 3) child-centered support materials mailed to participating families. The study will include an intervention group and a delayed control group. Feasibility of the digital intervention will be assessed at post-test only by recruitment, retention, usability, and acceptability. Implementation outcomes include measures of digital engagement, enactment, and intention to sustain, and will be collected at post-test only. Theoretical mediators include parent self-efficacy and behavioral capability and will be collected pre- and post-test. Behavioral outcomes, also collected at pre- and post-test, include mindful parenting, parent-child feeding practices, and physical activity parenting practices. Study assessments for the theoretical mediators and behavioral outcomes will be collected at Baseline (Time 1, pre-intervention) and at Post-Test (Time 2, post-intervention) at the same time for both groups. No additional assessments will be collected for the delayed control group at the conclusion of implementation.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a preschool-aged child (3-5 years) with no disabilities or conditions that impact typical eating and activity behaviors.
* Adult participants must have access to a smartphone, reliable internet at home, and can make video calls.

Exclusion Criteria:

* Adults who do not have a child aged 3-5 or child has a disability/condition that impact typical eating and activity behaviors.
* Technology access is limited.
* Adults who read, write or speak a language other than English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment | Baseline (week 0)
  Number of completed interest forms resulting in enrollment.
Retention | 10 weeks
  Proportion of intervention activities (e.g., app modules and assessments) completed.
Usability | Post-Intervention (week10)
  Mean scores using the System Usability Scale (SUS) to estimate ease of use, complexity, confidence in using, and likelihood of use (scale 0-5, with higher scores indicating higher rankings of usability)
Acceptability | 10 weeks
  Mean ratings of information helpfulness, goal setting, liking of the program, willingness to recommend, and desire for additional information (scale 0-5, with higher scores indicating higher acceptibility)
Digital Engagement | Post-Intervention (week10)
  Percentage of participants engaging with the app (i.e., engagement by topic, features, and temporal patterns), and by dosage (i.e., completion rates of modules and within-app activities).
Intention to sustain | Post-intervention (week 10)
  Qualitatively capture, via individual interviews, intervention strategies relating to target behaviors which were implemented or adopted.

SECONDARY OUTCOMES:
Mindful Parenting | Baseline (week 0) and Post-Intevention (week 10)
  Mean scores using the Interpersonal Mindfulness in Parenting survey (I-MP) will assess five constructs of mindful parenting: parent/caregiver listening with full attention, emotional awareness of self and child, self-regulation, compassion of self and child, non-judgmental acceptance of self and child). Scale, 0-5, with higher scores indicating higher mindful parenting.
Parent-Child Feeding Practices | Baseline (week 0) and Post-Intervention (week 10)
  Mean scores from the Food Parenting Inventory (FPI) will assess Autonomy (encourages exploration of new foods, offers new foods, repeatedly presents new foods) and Control (pressure to eat, food as reward). Scale, 0-5, with higher scores indicating more positive child feeding practices.
Physical Activity Parenting Practices | Baseline (week 0) and Post-Intervention (week 10)
  Mean scores from teh PA Parenting Practices (PAPP) will assess three parenting domains: Structure (nondirective support, supportive expectation, restriction of physical activity inside), Autonomy (autonomy support, guided choice), and Control (coercive control). Scale, 0-5, with higher scores indicating more positive PA practices.
Perceived Parenting Self-Efficacy | Baseline (week 0) and Post-Intervention (week 10)
  Mean scores of questions adapted from the Generalized Self-Efficacy Scales and will assess the offering of healthy foods, providing physical activity opportunities for their child, and engaging in positive interactions with their child related to healthy eating, physical activity, and modifying the home environment. Scale, 0-5, with higher scores indicating higher self-efficacy.
Behavioral capability skills | 10 weeks
  Means scores of questions adapted from the Feeding Knowledge Questionnaire to assess parent feeding knowledge and misconceptions, and the PLAYshop instrument adapted for use in parents of preschool-age children to assess physical literacy knowledge and confidence. Scale, 0-5, with higher scores indicating more higher behavioral capability.

OTHER OUTCOMES:
Child Meal Quality (exploratory) | Baseline (week 0) and Post-Intervention (week 10)
  Measured via food photography, meal quality will be assessed using Healthy Meal Index adequacy score (mean of 3 meals, range 0-55).
Child Meal Quantity (exploratory) | Baseline (week 0) and Post-Intervention (week 10)
  Measured via food photography, meal quantity will be determined by visual estimation of serving sizes (e.g., 1/4 c.)
Child's Dietary Intake (exploratory) | Baseline (week 0) and Post-Intervention (week 10)
  Mean scores of children's consumption of foods will be collected using the Dietary Screener Questionnaire (DSQ). Quantitative estimates of food and nutrient intake (e.g., cups of fruit, vegetables and ounce equivalents of whole grains). These quantitative estimates will be compared to recommended serving sizes from the Dietary Guidelines of Americans to determine if consumption of food groups is meeting, above or below guidelines.
Child Fundamental movement skill performance (exploratory) | Baseline (week 0) and Post-Intervention (week 10)
  Mean scores for objective control and locomotor skills will be assessed using Test for Gross Motor Development, 2nd Ed (TGMD-2) scoring protocol. Each skill is scored on a scale of 0-1 with subscale ranges of 0-6 for locomotor skills and 0-5 for object control skills.
Child Physical Activity Opportunities (exploratory) | Baseline (week 0) and Post-Intervention (week 10)
  Mean scores of opportunities for structured and unstructured PA will be assessed (scale, 0-5, with higher scores indicating more positive opportunities).
Home Food Environment (exploratory) | Baseline (week 0) and Post-Intervention (week 10)
  Frequency of the availability of Fruit, Convenience Foods, Beverages and Whole Grains; Physical activity equipment will be assessed via the HomeIDEAv3 instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Laura L Bellows, PhD, Principal Investigator — Cornell University
Locations (1):
- Cornell University, Ithaca, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Any unique resources will be made available immediately after publication. Procedures to protect the privacy of health data of individuals will be implemented to ensure HIPPA privacy standards are met. After the publication of outcome data, it will be made available to individuals who have IRB approval. The final dataset will be de-identified prior to sharing.
  We will insure that data and associated documentation is available to users only under a data sharing agreement that states a commitment to: 1) using the data only for research purposes, 2) securing the data using appropriate technology protection; and 3) destroying the data after analyses are completed.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication
Access Criteria: After the publication of outcome data, data will be made available to individuals who have IRB approval.

REFERENCES:
- [Background] Bellows LL, Oke S, Reyes LI, Carmona BA, Johnson SL. Development of a Digital Parent Intervention to Promote Healthy Eating and Activity in Preschoolers: The eHEROs Study. J Nutr Educ Behav. 2025 May;57(5):450-459. doi: 10.1016/j.jneb.2025.01.008. Epub 2025 Feb 7. PMID 39918513
- See also: Related Info — https://blogs.cornell.edu/healthbehavlab/know-how-program/

DOCUMENTS (1):
  • Study Protocol (2025-01-06): https://cdn.clinicaltrials.gov/large-docs/12/NCT07224412/Prot_000.pdf